CLINICAL TRIAL: NCT05887349
Title: Investigation of the Efficacy of Rocabado Exercises in Individuals With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: chronic neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The patients in the control group will be given cervical stabilization exercises consisting of 3 levels and increasing difficulty. The exercises will be taught to the patients level by level by the physiotherapist for 6 weeks. The subjects will perform the exercises for a total of 6 weeks. Before each exercise session, stretching exercises will be performed on the subjects.
  Interventions: Other: Neck Stabilization Exercise
- Intervention group (Experimental): The exercises to be applied to the control group for 6 weeks will be given to the intervention group in the same order and at weekly intervals. Additionally, Robacado exercises (jaw exercises) will be given to the individuals in this group.
  Interventions: Other: Neck Stabilization Exercise + Rocabado Exercises

INTERVENTIONS:
Other: Neck Stabilization Exercise — 1. Control Group exercise program (Cervical Stabilization exercises group)
  The patients in the control group will be given cervical stabilization exercises consisting of 3 levels and increasing difficulty. The exercises will be taught to the patients level by level by the physiotherapist for 6 weeks. The subjects will perform the exercises for a total of 6 weeks. Before each exercise session, stretching exercises will be performed on the subjects.
  Arms: Control Group
Other: Neck Stabilization Exercise + Rocabado Exercises — 2. Intervention group exercise program (the group to which Robacado exercises will be added in addition to cervical stabilization exercises) The exercises to be applied to the control group for 6 weeks will be given to the intervention group in the same order and at weekly intervals. In addition, individuals in this group will be given Robacado exercises.
  Robacado exercises:
  1. Resting position for the tongue: The tip of the tongue is placed on the upper palate, just behind the front teeth (resting position for the tongue).
  2. When the body is in an upright position, scapular retraction and depression movements are performed without disturbing the position of the cervical region.
  3. When the body is in an upright position, at C2-C7 levels, hands are clamped on the neck and cranio-cervical flexion is studied.
  Arms: Intervention group

SUMMARY:
Nerve compression, disc herniation, and fracture-related factors may play a role in the etiology of chronic neck pain, or the pain may not be associated with a specific cause. In the cervical region, muscles, fascia, disc, nerve root and facet joints are the structures that carry pain. Problems related to these structures can also cause pain in the cervical region and shoulder, arm, interscapular region and craniocervical structures. The stomatognathic system is the integrity of the structures that perform the functions of chewing, swallowing and speaking. This system in the head and neck region; It consists of bones, muscles, joints, ligaments, teeth, supporting dental tissues, glands, tongue, mouth and surrounding tissues, and neuromuscular system. The relationship between the stomatognathic and craniocervical systems is demonstrated by the interaction between masticatory and cervical muscles. Wiesinger et al. examined the relationship between spinal pain and temporamandibular joint disorders in a large sample and stated that both conditions may share common risk factors or affect each other. The coexistence of cervical spine and temporomandibular joint pathologies (TMJ) is explained by the neuroanatomical convergence of nociceptive neurons receiving trigeminal and neck sensory inputs. Studies have shown that neck disability may be accompanied by jaw joint disability, masseter myofascial pain, and regional muscle tenderness. Olivio et al. He reported that the treatment of individuals with TMJ pathology should also focus on the neck region, because improvement of one may affect the other. Based on this idea, Calixtre et al. reported that they achieved positive improvements in pain and jaw functions in their study investigating the effects of cervical region mobilization and exercises on individuals with TMJ.

DETAILED DESCRIPTION:
Nerve compression, disc herniation, and fracture-related factors may play a role in the etiology of chronic neck pain, or the pain may not be associated with a specific cause. In the cervical region, muscles, fascia, disc, nerve root and facet joints are the structures that carry pain. Problems related to these structures can also cause pain in the cervical region and shoulder, arm, interscapular region and craniocervical structures. The stomatognathic system is the integrity of the structures that perform the functions of chewing, swallowing and speaking. This system in the head and neck region; It consists of bones, muscles, joints, ligaments, teeth, supporting dental tissues, glands, tongue, mouth and surrounding tissues, and neuromuscular system. The relationship between the stomatognathic and craniocervical systems is demonstrated by the interaction between masticatory and cervical muscles. Wiesinger et al. examined the relationship between spinal pain and temporamandibular joint disorders in a large sample and stated that both conditions may share common risk factors or affect each other. The coexistence of cervical spine and temporomandibular joint pathologies (TMJ) is explained by the neuroanatomical convergence of nociceptive neurons receiving trigeminal and neck sensory inputs. Studies have shown that neck disability may be accompanied by jaw joint disability, masseter myofascial pain, and regional muscle tenderness. Olivio et al. He reported that the treatment of individuals with TMJ pathology should also focus on the neck region, because improvement of one may affect the other. Based on this idea, Calixtre et al. reported that they achieved positive improvements in pain and jaw functions in their study investigating the effects of cervical region mobilization and exercises on individuals with TMJ.

In the treatment of chronic neck pain, it has been shown that craniocervical flexion exercise, cervical stabilization and endurance exercises, aerobic exercises, proprioceptive exercises and patient education, especially strengthening exercises for deep and superficial flexor muscles, reduce pain and improve quality of life by increasing muscle strength and functions. In the literature, the number of studies investigating the effectiveness of an exercise program for the jaw joint in individuals with chronic neck pain is quite limited. In this context, our aim is to investigate the effects of Rocabado exercises, one of the jaw joint exercises, on pain, pain threshold/tolerance, range of motion, proprioception, disability, quality of life, muscle strength, muscle endurance, sleep quality and posture in individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having neck pain for 3 months,
* Being sedentary
* Not participating in any physical therapy program in the last 6 months.

Exclusion Criteria:

* Being history of previous spinal surgery or trauma,
* Beingneurological deficit, vestibular pathology, neurological, cardiopulmonary, musculoskeletal problems affecting physical performance
* Being any pathology in the shoulder joint, any pathology in the jaw joint, and pregnancy were determined.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Disability level | 6 week
  Neck disability caused by neck pain was evaluated with the Neck Disability Index (NDI), which has been validated and reliable in Turkish. NDI was developed to evaluate the impact of neck pain on daily life activities (pain intensity, personal care, lifting, reading, concentration, work, driving, sleep and leisure activities) and consists of 10 sections. Each section is scored between 0 and 5 points. The total score obtained is between 0-50. Scores between 0-4 indicate no disability, scores between 5-14 indicate mild disability, scores between 15-24 indicate moderate disability, scores between 25-34 indicate severe disability, and scores above 35 indicate full disability.

SECONDARY OUTCOMES:
Joint Range of Motion assessment | 6 week
  Cervical region flexion, extension, right-left rotation and right-left lateral flexion range of motion of individuals will be evaluated with clinical goniometer.
Pain assessment | 6 week
  Visual Analog Scale (VAS) will be used for the presence and severity of neck pain in the individuals included in the study. Each participant will be asked about the presence and severity of pain at the beginning and end of the study and recorded. For VAS, individuals are asked to indicate the degree of pain they have on the VAS scale, numbered from 0 to 10 on a straight line, with "0" being no pain and "10" being the most severe pain and recorded.
Proprioception assessment | 6 week
  The Cervical Joint Position Error Test (CJPET) is used to evaluate cervical region proprioception. CJPET assesses cervical proprioception in four positions (flexion, extension, left rotation, and right rotation). It is based on the principle of finding a point while the eyes are closed. 10 repetitions for each position were done. The first four measurements are trials and the average of the last six measurements gives us the joint position error
Balance | 6 week
  Participants' static and dynamic balance was assessed using the Biodex balance system (Biodex, Inc., Shirley, New York). The device consists of a mobile balance platform that provides quantitative measurements of postural control in the sagittal and frontal planes in a 360° arc of motion up to 20° surface inclination. The device evaluates anterior-posterior stability index (A-P), medial-lateral stability index (M-L), and overall stability index (overall variance in both planes).
Muscle endurance | 6 week
  The endurance of the cervical region flexor muscles was evaluated in the supine position, with the hands next to the body and in the hook position. Participants were asked to gently bring their chin closer to the chest area. The time it remained in this position was recorded in seconds. The evaluator placed his hand under the occiput to determine whether the position was maintained. The endurance of the cervical region extensor muscles was evaluated while the participant was in the prone position. The participant's head was positioned so that it hung over the bed and a 2 kg weight bag was tied to its head. The time he maintained this position was recorded in seconds.
Pain threshold and tolerance | 6 week
  Participants' pain threshold and tolerance to pressure were evaluated using a digital algometer device (JTech Medical Industries, ZEVEX Company). It is stated that the reliability of this digital algometer is high. In the evaluation of pain threshold and tolerance, the midpoint of the upper part of the trapezius muscle between the 7th cervical vertebra and the acromion was taken as a reference. Evaluations were made with a 1 cm2 disc head apparatus connected to the algometer device that gives results in kg/cm2.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No